CLINICAL TRIAL: NCT06148805
Title: Effect of Pilates Exercises and Diaphragm Manual Therapy Techniques in Rotator Cuff Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Samir Ismail El shahawy, principal investigator mona samir ismail el shahawy, Prof.Adel Rashad Ahmed, prof.Amaal Hassan Ibrahim, clinical Dr.Mohamed Ali Amin, asst. profGhada Abed Elmoniem Abed Allaha, Ministry of Health and Population, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004001
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Shoulder Tendinitis; Shoulder Rotator Cuff Tendinopathy
Keywords: Shoulder Tendinitis; shoulder rotator cuff tendinopathy; Pilates exercise; diaphragmatic respiratory technique; physical therapy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: 1. Patients diagnosed with rotator cuff tendinopathy for duration greater than three months (Eda and Emin,2016).
  2. 40 and 60 years of age from both genders (Yamamoto et al.,2019)
  3. Patient's BMI within normal range between 18.5 and 24.9 (Gumina et al.,2014)
  4. patients complain of shoulder pain at the tip of the shoulder and the upper, outer arm. The pain is aggravated by reaching, pushing, pulling, lifting, positioning the arm above the shoulder level, or lying on the side (Stiphen and Micheal,1021).
  5. The arm pain during resisted testing (usually abduction and/or lateral rotation) (Eda and Emin,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pilates Group (Experimental): fifteen patients diagnosed with shoulder rotator cuff tendinopathy for at least 3 months randomly selected from ministry of health units will receive Pilates exercises program additional to traditional (RCT) physical therapy program containing Hot-Pack (HP), Therapeutic Ultrasound (US) and upper extremity strengthening and stretching exercise program)
  * The assessment of pain intensity was carried out by visual analog scale
  * The assessment of pain threshold was carried out by pressure algometer.
  * The assessment of lateral rotation strength and abduction strength were carried out by hand heled dynamometer.
  * The assessment of shoulder function was carried out by Arabic version of the Disability of the Arm, Shoulder and Hand (DASH-Arabic)
  * The assessment of the functional exercise performance was carried out by Six-min walk test
  Interventions: Other: pilates exercise and diaphragm manual technique
- diaphragmatic Group (Experimental): fifteen patients diagnosed with shoulder rotator cuff tendinopathy for at least 3 months randomly selected from ministry of health units will receive diaphragm manual therapy techniques and traditional rotator cuff tendinopathy physical therapy program containing Hot-Pack (HP), Therapeutic Ultrasound (US) and upper extremity strengthening and stretching exercise program)
  * The assessment of pain intensity was carried out by visual analog scale
  * The assessment of pain threshold was carried out by pressure algometer.
  * The assessment of lateral rotation strength and abduction strength were carried out by hand heled dynamometer.
  * The assessment of shoulder function was carried out by Arabic version of the Disability of the Arm, Shoulder and Hand (DASH-Arabic)
  * The assessment of the functional exercise performance was carried out by Six-min walk test
  Interventions: Other: pilates exercise and diaphragm manual technique
- traditional Group (Active Comparator): fifteen patients diagnosed with shoulder rotator cuff tendinopathy for at least 3 months randomly selected from ministry of health units will receive 15 received traditional rotator cuff tendinopathy physical therapy program containing Hot-Pack (HP), Therapeutic Ultrasound (US) and upper extremity strengthening and stretching exercise program)
  * The assessment of pain intensity was carried out by visual analog scale
  * The assessment of pain threshold was carried out by pressure algometer.
  * The assessment of lateral rotation strength and abduction strength were carried out by hand heled dynamometer.
  * The assessment of shoulder function was carried out by Arabic version of the Disability of the Arm, Shoulder and Hand (DASH-Arabic)
  * The assessment of the functional exercise performance was carried out by Six-min walk test
  Interventions: Other: pilates exercise and diaphragm manual technique
- pilates and diaphragmatic Group (Experimental): fifteen patients diagnosed with shoulder rotator cuff tendinopathy for at least 3 months randomly selected from ministry of health units will receive diaphragm manual therapy, Pilates exercises program and traditional rotator cuff tendinopathy physical therapy program containing Hot-Pack (HP), Therapeutic Ultrasound (US) and upper extremity strengthening and stretching exercise program)
  * The assessment of pain intensity was carried out by visual analog scale
  * The assessment of pain threshold was carried out by pressure algometer.
  * The assessment of lateral rotation strength and abduction strength were carried out by hand heled dynamometer.
  * The assessment of shoulder function was carried out by Arabic version of the Disability of the Arm, Shoulder and Hand (DASH-Arabic)
  * The assessment of the functional exercise performance was carried out by Six-min walk test
  Interventions: Other: pilates exercise and diaphragm manual technique

INTERVENTIONS:
Other: pilates exercise and diaphragm manual technique — pilates exercises
  Other Names: exercises

SUMMARY:
1. To investigate the effect of Pilates exercises program on pain intensity, pain threshold, shoulder lateral rotator strength, abduction strength and shoulder function in patients with (RCT).
2. To investigate the effect of diaphragm manual therapy techniques on pain intensity, pain threshold, shoulder lateral rotator strength, abduction strength and shoulder function in patients with (RCT).
3. To determine the effect of combination between Pilates exercises program and diaphragm manual therapy techniques on pain intensity, pain threshold, shoulder lateral rotator strength, abduction strength and shoulder function in patients with (RCT).

DETAILED DESCRIPTION:
Musculoskeletal complains are common work-related problems in Egypt. Egyptian preparatory school teachers were 96%. Dental society revealed high response rate (93%) with 53.8% have complains related to neck/shoulder .Physical therapists (PTs) are frequently exposed to work-related musculoskeletal disorders .Shoulder problems represent (47.7%).Printing workers and municipal solid waste collectors are another group having high prevalence of work-related musculoskeletal disorders that might be related to some individual factors (age, BMI, and duration of employment).

Since pilates shoulder exercise influence shoulder function and pain and to considering the relationship between shoulder muscles and the thoracic cage expansion. Consequently, it is worthy to investigate the efficacy of Pilates exercises program with diaphragm manual therapy techniques in pain intensity, pain threshold, shoulder lateral rotator strength, abduction strength and shoulder function on patient with rotator cuff tendinopathy aiming for function improvement and pain decrease. Therefore, this study is being conducted for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with rotator cuff tendinopathy for duration greater than three months
2. Body Mass Index between 18.5 and 24.9
3. patients complain of shoulder pain at the tip of the shoulder and the upper, outer arm.
4. pain during resisted arm test (usually abduction and/or lateral rotation) (

Exclusion Criteria:

* 1. shoulder stiffness 2. Previous dislocation or sublation of shoulder joint. 3. Previous shoulder surgery 4. Glenohumeral joint and acromioclavicular joint degeneration 5. Neurological deficit in the neck or arm 6. Heavy Smokers. 7. Any Cardiopulmonary pathology. 8. Recent Thoracic surgery 9. Any deformity of spine 10. History of Thyroid Disorders 11. Cognitive impairment

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
shoulder pain | 4 weeks
  visual analog scale (scale from 0 to 10 where 0 means no pain and 10 means unbearable pain pain threshold will be carried out by pressure algometer
strength of shoulder muscle | 4 weeks
  hand heled dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ali, professor, Study Director — Ministry of Health
Locations (1):
- MOH, Cairo, Ramsis Saint Abbassia , Cairo., Egypt

IPD SHARING:
Plan to Share IPD: No